CLINICAL TRIAL: NCT04059666
Title: Gastrointestinal Tract Microbiome in Healthy Term Infants Receiving Mother'S-own Breast Milk or Cow's Milk-based Infant Formulas
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrolment
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 3390-1
Record Dates: First submitted 2019-05-08; First posted 2019-08-16 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Gastrointestinal Microbiome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator)
  Interventions: Other: Control
- Investigational (Experimental)
  Interventions: Other: Investigational
- Mother's-own Breast Milk (No Intervention)

INTERVENTIONS:
Other: Investigational — Cow's milk-based Infant Formula with whey protein-lipid concentrate
  Arms: Investigational
Other: Control — Cow's milk-based Infant Formula
  Arms: Control

SUMMARY:
This clinical trial will compare stool and oral microbiome composition between infants fed breast milk or one of two infant formulas for a 60 day feeding period.

ELIGIBILITY:
Inclusion Criteria:

* 7-18 days of age at Visit 1
* Singleton birth
* Gestational age of 37-42 weeks
* Birth weight of 2500 g (5 lbs 8 oz) or more
* Parent or legal guardian agrees not to enroll infant in another interventional clinical study while participating in this study
* Signed informed consent and use of PHI for infant and birth mother
* Receipt of three protocol-compliant Baseline stool samples

Infants receiving formula:

* Exclusively receiving infant formula for at least 24 hours prior to randomization
* Parent(s) or legal guardian has full intention to exclusively feed study formula during the study period

Infants receiving human milk:

* Mother has intention to exclusively provide mother's-own breast milk for the duration of the study

Exclusion Criteria:

* Caesarean delivery
* Infant consumption of donor milk prior to randomization/registration
* Maternal antibiotic use within 48 hours prior to or at time of delivery
* Maternal antibiotic use while providing mother's-own breast milk to infant
* Infant use of systemic antibiotics prior to randomization/registration
* Any signs of an acute infection (i.e. fever, diarrhea) at randomization/registration
* Weight at Visit 1 is <95% of birth weight
* Infant use of probiotics
* Evidence of significant feeding difficulties
* Infant was born large for gestational age
* History of underlying metabolic or chronic disease or congenital malformation
* Infant is immunocompromised

Infants receiving human milk:

* Consumption of infant formula from 1 day of age

Ages: 7 Days to 18 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Comparison of stool microbiome between breast fed and formula fed babies | Over 60 days
  Stool collection

SECONDARY OUTCOMES:
Oral microbiome at each visit | Over 60 days
  Buccal swab
Stool molecules at each visit | Over 60 days
  Stool sample
24 hour recall of formula intake | 2 times over 60 days
  24 hour recall questionnaire
Stool color and consistency | 3 times over 60 days
  Color and consistency
Medically confirmed adverse events | 60 days
  Medically confirmed adverse events
Stool pH | Over 60 days
  pH

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Birmingham Pediatric Associates, Birmingham, Alabama
  - Children's Research, LLC, Altamonte Springs, Florida
  - Owensboro Pediatrics, Owensboro, Kentucky
  - Holston Medical Group, Kingsport, Tennessee
  - Memphis & Shelby County Pediatric, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christensen C, Kok CR, Harris CL, Moore N, Wampler JL, Zhuang W, Wu SS, Hutkins R, Izard J, Auchtung JM. Microbiota, metabolic profiles and immune biomarkers in infants receiving formula with added bovine milk fat globule membrane: a randomized, controlled trial. Front Nutr. 2024 Oct 4;11:1465174. doi: 10.3389/fnut.2024.1465174. eCollection 2024. PMID 39444571